CLINICAL TRIAL: NCT02455401
Title: Effect of Remifentanil on Postoperative Vomiting in Children Undergoing Strabismus Surgery During Sevoflurane Anesthesia
Brief Title: Effect of Remifentanil on Postoperative Vomiting in Pediatric Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant Professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2015-024
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Strabismus
Keywords: Postoperative Vomiting
MeSH Terms: conditions — Strabismus; Postoperative Nausea and Vomiting | interventions — Remifentanil; halofantrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- high dose remifentanil group (Experimental): Intervention: high dose remifentanil will be administrated.
  Interventions: Drug: High dose remifentanil
- low dose remifentanil group (Experimental): Intervention: low dose remifentanil will be administrated
  Interventions: Drug: Low dose remifentanil
- No remifentanil group (Placebo Comparator): Intervention: no remifenatnil will be administrated
  Interventions: Drug: No remifentanil

INTERVENTIONS:
Drug: High dose remifentanil — Intervention: continuously intravenous infusion of remifentanil 0.1 mcg/kg/min after bolus injection of remifentanil 1.0 mcg/kg for 2 minutes
  Other Names: High dose remifentanil (Ultiva,Glaxosmithkline, UK)
  Arms: high dose remifentanil group
Drug: Low dose remifentanil — Intervention: continuously intravenous infusion of remifentanil 0.1 mcg/kg/min after bolus injection of remifentanil 0.5 mcg/kg for 2 minutes
  Other Names: Low dose remifentanil (Ultiva, Glaxosmithkline, UK)
  Arms: low dose remifentanil group
Drug: No remifentanil — Intervention: no remifentanil will be administrated
  Other Names: No remifentanil (Ultiva, Glaxosmithkline, UK)
  Arms: No remifentanil group

SUMMARY:
The purpose of this study is to compare the effect of remifentanil on postoperative vomiting in children undergoing strabismus surgery during sevoflurane anesthesia.

DETAILED DESCRIPTION:
Children undergoing strabismus surgery frequently experience postoperative vomiting (POV) that results in dehydration, aspiration pneumonia, bleeding, delayed hospital discharge, as well as decreased parental satisfaction and an unpleasant experience for the pediatric patients. Although administration of perioperative opioids increases POV incidence, remifentanil has less affect the incidence of POV than other opioids such as fentanyl. However, there are few study that evaluate the effects of remifentanil on the incidence of POV. Therefore, the investigators will conducted the study that the effects of remifentanil on the incidence of POV in children undergoing strabismus surgery during sevoflurane anesthesia. One hundred five children from 3 to 6 yr of age, ASA physical status 1 or 2 were assigned randomly selected to one of three groups: high dose remifentanil group (bolus 1.0 mcg/kg; infusion 0.1 mcg/kg/min), low remifentanil group (bolus 0.5 mcg/kg; infusion 0.1 mcg/kg/min), or no remifentanil group (no remifentanil administration). Primary endpoint, the incidence of POV for 24 hours postoperatively, will be compared between three study groups.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing elective strabismus surgery under sevoflurane anesthesia

Exclusion Criteria:

* children who experienced postoperative retching or vomiting
* children who have taken anti-emetic medications within 24 hours before surgery
* children who experienced motion sickness

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative vomiting in PACU and surgical ward | from extubation to 24 hours
  Vomiting is expulsion of gastric contents. Incidence of vomiting will be compared between the groups.

SECONDARY OUTCOMES:
postoperative pain in PACU and surgical ward | from extubation to 24 hours
  Postoperative pain will be assessed using Faces Pain Rating Scale.
postoperative emergence agitation | from extubation to 24 hours
  Postoperative emergence agitation will be assessed using Pediatric Anesthesia Emergence Delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Lee, M.D., Principal Investigator — Inje University
Locations (1):
- Haeundae paik hospital, inje university, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No